CLINICAL TRIAL: NCT02415842
Title: An Exploratory, Retrospective Laboratory Evaluation of the Humoral Immune Response in Adults and Children to the H1 HA Stalk Domain and Other Influenza A Virus Protein Epitopes, After Administration of GSK Biologicals' Pandemic Influenza Vaccines
Brief Title: A Laboratory Evaluation of the Humoral Immune Response in Adults and Children to the H1 Hemagglutinin (HA) Stalk Domain and Other Influenza A Virus Protein Epitopes, After Administration of GlaxoSmithKline (GSK) Biologicals' Pandemic Influenza Vaccines
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 201598
Record Dates: First submitted 2015-03-26; First posted 2015-04-14 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Immunologic Tests
Keywords: Supra-seasonal influenza vaccine; Pandemic; Exploratory; Protein epitopes; Laboratory evaluation; Retrospective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum samples

GROUPS / COHORTS (13):
- H1N1_AS Group: Subjects 19-40 years of age (in H1N1 cohort of primary completed study Q-PAN H1N1-019 (113536) (A/California/07/2009)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21 and TIV at Day 42.
  Interventions: Other: Serum samples
- H1N1_NAS Group: Subjects 19-40 years of age (in H1N1 cohort of primary completed study -Q-PAN H1N1-019 (113536) (A/California/07/2009)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21 and TIV at Day 42
  Interventions: Other: Serum samples
- H5N1_AS Group: Subjects 18-49 years of age (in H5N1 cohort of primary completed study CC-PAN H5N1-001 (114371)(A/Indonesia/5/2005 RG)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21
  Interventions: Other: Serum samples
- H5N1_NAS Group: Subjects 18-49 years of age (in H5N1 cohort of primary completed study CC-PAN H5N1-001 (114371)(A/Indonesia/5/2005 RG)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21.
  Interventions: Other: Serum samples
- H9N2_AS Group: Subjects 18-64 years of age (in H9N2 cohort of primary completed study Q-PAN H9N2-001 (116358) (A/chicken/Hong Kong/G9/1997 NIBRG-91)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21 and saline placebo at Day 182.
  Interventions: Other: Serum samples
- H9N2_NAS Group: Subjects 18-64 years of age (in H9N2 cohort of primary completed studyQ-PAN H9N2-001 (116358)(A/chicken/Hong Kong/G9/1997 NIBRG-91)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21 and with saline placebo at Day 182.
  Interventions: Other: Serum samples
- DQIV_NAS Group: Subjects 18-≤39 years of age (in D-QIV cohort of primary completed study FLU D-QIV-015 (201251) (A/Christchurch/16/2010 (H1N1)pdm09, A/Texas/50/2012 (H3N2), B/Massachusetts/02/2012, B/Brisbane/60/2008)) who were administered 15 µg HA (no AS) of each of 4 strains (total 60 µg HA) at Day 0.
  Interventions: Other: Serum samples
- QPAN_C Group: Subjects 18-40 years of age (in Q-PAN cohort of primary completed study Q-PAN-005 (110624)) who were administered 3.8 µg A/Indonesia/5/05 (H5N1) with AS03A on Day 0; phosphate buffer saline (PBS) preserved with 20 ppm thimerosal on Day 182; 3.8 µg A/turkey/Turkey/1/05 (H5N1) with AS03A on Day 549.
  Interventions: Other: Serum samples
- QPAN5_G Group: Subjects 18-40 years of age (in Q-PAN cohort of primary completed study Q-PAN-005 (110624)) who were administered PBS preserved with 20 ppm thimerosal on Day 0; 3.8 µg A/turkey/Turkey/1/05 (H5N1) with AS03A on Days 182 and 549.
  Interventions: Other: Serum samples
- H5N1_VT Group: Subjects 18-60 years of age (in H5N1 cohort of primary completed study H5N1-012 (107495) A/Vietnam/1194/2004-like or A/Indonesia/05/2005-like) who received two administrations of the adjuvanted (AS03A) pandemic influenza vaccine (3.8 µg) containing the Vietnam (VT) strain at Day 0 and Month 12.
  Interventions: Other: Serum samples
- H5N1_IN Group: Subjects 18-60 years of age (in H5N1 cohort of primary completed studyH5N1-012 (107495) A/Vietnam/1194/2004-like or A/Indonesia/05/2005-like) who received one administration(3.8 µg) of the adjuvanted (AS03A) pandemic influenza vaccine containing the Vietnam (VT) strain at Day 0 and one administration(3.8 µg) of the adjuvanted (AS03A) pandemic vaccine containing the Indonesia (IN) strain at Month 12.
  Interventions: Other: Serum samples
- H5N1_PAS Group: Subjects 6-35 months of age (in H5N1 cohort of primary completed study Q-PAN H5N1-AS03-021 (114464)(A/Indonesia/5/2005 RG)) who were administered adjuvanted (AS03B) pandemic vaccine with 1.9 µg HA (hemagglutinin) at Days 0 and 21.
  Interventions: Other: Serum samples
- H5N1_PCN Group: Subjects 6-35 months of age (in H5N1 cohort of primary completed study Q-PAN H5N1-AS03-021 (114464)(A/Indonesia/5/2005 RG)) who were administered placebo at Days 0 and 21.
  Interventions: Other: Serum samples

INTERVENTIONS:
Other: Serum samples — The archived sera samples collected in previously completed pandemic influenza vaccine clinical trials (H1N1, H5N1, and H9N2 pandemic vaccines in adult trials and H5N1 pandemic vaccine in a pediatric trial) will be tested in this study.

SUMMARY:
The purpose of this exploratory, retrospective laboratory study is to assess the humoral immune response to H1 hemagglutinin stalk domain and other influenza A virus protein epitopes following administration, in adults and children, of GSK Biologicals' adjuvanted and unadjuvanted pandemic influenza vaccines, using archived serum samples from previously completed clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Not applicable since no subjects will be actively enrolled in this study; only the sera samples of the subjects who were a part of previously conducted primary trials will be used for testing. However, the archived serum samples of only those subjects who satisfy the following criteria will be included in this study:

* Subjects who received two doses of influenza vaccine 21 days apart and were included in the ATP cohort for immunogenicity and Persistence cohort (depending on the study) in the primary studies listed.
* Subjects who had agreed that their blood samples could be used for further research while giving informed consent for any of the primary studies listed.
* Subjects who have sufficient residual sample volume (i.e., ≥0.5 mL) of serum at all time points.
* Subjects with vaccine homologous neutralizing antibody result available at Day 0 and at 21 (25 samples available per group in Study H9N2-001)

Exclusion Criteria:

* Not applicable since no subjects will be actively enrolled in this study; only the serum samples of the subjects who were a part of previously conducted trials will be used for testing.

Ages: 6 Months to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Archived serum samples to be evaluated in this study were collected from adults 18-64 years of age and children 6-35 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nachbagauer R, Salaun B, Stadlbauer D, Behzadi MA, Friel D, Rajabhathor A, Choi A, Albrecht RA, Debois M, Garcia-Sastre A, Rouxel RN, Sun W, Palese P, Mallett CP, Innis BL, Krammer F, Claeys C. Pandemic influenza virus vaccines boost hemagglutinin stalk-specific antibody responses in primed adult and pediatric cohorts. NPJ Vaccines. 2019 Dec 6;4:51. doi: 10.1038/s41541-019-0147-z. eCollection 2019. PMID 31839997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects analyzed in this study were subjects enrolled and analyzed in the According-to-Protocol (ATP)cohort for immunogenicity from Hemagglutinin (HA) Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines).
Pre-assignment Details: The HA Group 1-related studies were the followings: (FLU Q-PAN H1N1-019; [113536]; FLU CC-PAN H5N1-001[114371]; FLU Q-PAN H9N2-001[116358]; FLU Q-PAN-005[110624]; H5N1-012[107495]; FLU D-QIV-015[201251] and FLU Q-PAN H5N1-AS03-021[114464]).
Groups:
- H1N1_AS: Subjects 19-40 years of age (in H1N1 cohort of primary completed study Q-PAN H1N1-019 (113536) (A/California/07/2009)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21 and TIV at Day 42
- H1N1_NAS: Subjects 19-40 years of age (in H1N1 cohort of primary completed study -Q-PAN H1N1-019 (113536) (A/California/07/2009)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21 and TIV at Day 42
- H5N1_AS: Subjects 18-49 years of age (in H5N1 cohort of primary completed study CC-PAN H5N1-001 (114371)(A/Indonesia/5/2005 RG)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21
- H5N1_NAS: Subjects 18-49 years of age (in H5N1 cohort of primary completed study CC-PAN H5N1-001 (114371)(A/Indonesia/5/2005 RG)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21
- H9N2_AS: Subjects 18-64 years of age (in H9N2 cohort of primary completed study Q-PAN H9N2-001 (116358) (A/chicken/Hong Kong/G9/1997 NIBRG-91)) who were administered adjuvanted (AS03A) pandemic vaccine with 3.75 µg HA (hemagglutinin) at Days 0 and 21 and saline placebo at Day 182.
- H9N2_NAS: Subjects 18-64 years of age (in H9N2 cohort of primary completed studyQ-PAN H9N2-001 (116358)(A/chicken/Hong Kong/G9/1997 NIBRG-91)) who were administered unadjuvanted pandemic vaccine with 15 µg HA (hemagglutinin) at Days 0 and 21 and with saline placebo at Day 182.
- DQIV_NAS: Subjects 18-≤39 years of age (in D-QIV cohort of primary completed study FLU D-QIV-015 (201251) (A/Christchurch/16/2010 (H1N1)pdm09, A/Texas/50/2012 (H3N2), B/Massachusetts/02/2012, B/Brisbane/60/2008)) who were administered 15 µg HA (no AS) of each of 4 strains (total 60 µg HA) at Day 0.
- QPAN5_C: Subjects 18-40 years of age (in Q-PAN cohort of primary completed study Q-PAN-005 (110624)) who were administered 3.8 µg A/Indonesia/5/05 (H5N1) with AS03A on Day 0; phosphate buffer saline (PBS) preserved with 20 ppm thimerosal on Day 182; 3.8 µg A/turkey/Turkey/1/05 (H5N1) with AS03A on Day 549.
- QPAN5_G: Subjects 18-40 years of age (in Q-PAN cohort of primary completed study Q-PAN-005 (110624)) who were administered PBS preserved with 20 ppm thimerosal on Day 0; 3.8 µg A/turkey/Turkey/1/05 (H5N1) with AS03A on Days 182 and 549.
- H5N1_VT: Subjects 18-60 years of age (in H5N1 cohort of primary completed study H5N1-012 (107495) A/Vietnam/1194/2004-like or A/Indonesia/05/2005-like) who received two administrations of the adjuvanted (AS03A) pandemic influenza vaccine (3.8 µg) containing the Vietnam (VT) strain at Day 0 and Month 12.
- H5N1_IN: Subjects 18-60 years of age (in H5N1 cohort of primary completed studyH5N1-012 (107495) A/Vietnam/1194/2004-like or A/Indonesia/05/2005-like) who received one administration (3.8 µg) of the adjuvanted (AS03A) pandemic influenza vaccine containing the Vietnam (VT) strain at Day 0 and one administration (3.8 µg) of the adjuvanted (AS03A) pandemic vaccine containing the Indonesia (IN) strain at Month 12
- H5N1_PAS: Subjects 6-35 months of age (in H5N1 cohort of primary completed study Q-PAN H5N1-AS03-021 (114464)(A/Indonesia/5/2005 RG)) who were administered adjuvanted (AS03B) pandemic vaccine with 1.9 µg HA (hemagglutinin) at Days 0 and 21.
- H5N1_PCN: Subjects 6-35 months of age (in H5N1 cohort of primary completed study Q-PAN H5N1-AS03-021 (114464)(A/Indonesia/5/2005 RG)) who were administered placebo at Days 0 and 21.
Period: Overall Study
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS | DQIV_NAS | QPAN5_C | QPAN5_G | H5N1_VT | H5N1_IN | H5N1_PAS | H5N1_PCN
Started | 29 | 29 | 29 | 27 | 30 | 30 | 30 | 26 | 29 | 53 | 49 | 33 | 20
Completed | 29 | 29 | 29 | 27 | 30 | 30 | 30 | 26 | 29 | 53 | 49 | 33 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS | DQIV_NAS | QPAN5_C | QPAN5_G | H5N1_VT | H5N1_IN | H5N1_PAS | H5N1_PCN | Total
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30 | 30 | 26 | 29 | 53 | 49 | 33 | 20 | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 20 | 53
  Between 18 and 65 years | 29 | 29 | 29 | 27 | 30 | 30 | 30 | 26 | 29 | 53 | 49 | 0 | 0 | 361
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 17 | 18 | 14 | 16 | 22 | 12 | 16 | 21 | 28 | 16 | 10 | 227
  Male | 10 | 11 | 12 | 9 | 16 | 14 | 8 | 14 | 13 | 32 | 21 | 17 | 10 | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Hispanic or Latino | 2 | 1 | 5 | 4 | 2 | 2 | 0 | 3 | 4 | 0 | 0 | 3 | 0 | 26
  Not American Hispanic or Latino | 27 | 28 | 24 | 23 | 28 | 28 | 0 | 23 | 25 | 53 | 49 | 30 | 20 | 358
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 30
Age continuous-pediatric study [Mean (Standard Deviation); unit: Months] — Population: This category applies to H5N1_PAS and H5N1_PCN groups (pediatric groups). This category is not applicable to any of the adults groups.
  Months
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 20 | 53
    (all) |  |  |  |  |  |  |  |  |  |  |  | 22.6 (7.6) | 23.5 (6.9) | 22.9 (7.3)
Age continuous- adults subjects [Mean (Standard Deviation); unit: Years] — Population: This category applies to the adults groups. This category is not applicable to H5N1_PAS and H5N1_PCN groups (pediatric groups).
  Years
    number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30 | 30 | 26 | 29 | 53 | 49 | 0 | 0 | 361
    (all) | 28.5 (6.5) | 29.3 (6.8) | 30.4 (8.3) | 31.4 (9.1) | 43.3 (11.9) | 42.6 (13.6) | 26.7 (5.7) | 29.4 (6.5) | 29.6 (6.8) | 35.8 (12.1) | 35.4 (12.5) |  |  | 32.9 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Equal or Above the Cut-off of 66 EU/mL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from Hemagglutinin (HA) Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with concentrations greater or equal than 66 Elisa Unit per milliliter (EU/mL).
Time Frame: At Day 0 (Pre-vaccination), Day 21 (Post-vaccination 1), Day 42 (Post-vaccination 2), Day 182 (post-vaccination 2) and Day 385 (Post-vaccination 2 -for H5N1 cohorts only)
Population: All subjects from each study cohort with available results were included in the analysis for this study. All subjects selected were from the ATP cohort for immunogenicity of respective primary studies.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30
Percentage of subjects
  Day 0: number analyzed (Participants) | 27 | 25 | 29 | 27 | 30 | 30
  Day 0 | 100 [87.2 to 100] | 100 [86.3 to 100] | 100 [88.1 to 100] | 100 [87.2 to 100] | 100 [88.4 to 100] | 100 [88.4 to 100]
  Day 21: number analyzed (Participants) | 28 | 25 | 29 | 27 | 30 | 30
  Day 21 | 100 [87.7 to 100] | 100 [86.3 to 100] | 100 [88.1 to 100] | 100 [87.2 to 100] | 100 [88.4 to 100] | 100 [88.4 to 100]
  Day 42: number analyzed (Participants) | 27 | 27 | 29 | 27 | 30 | 30
  Day 42 | 100 [87.2 to 100] | 100 [87.2 to 100] | 100 [88.1 to 100] | 100 [87.2 to 100] | 100 [88.4 to 100] | 100 [88.4 to 100]
  Day 182: number analyzed (Participants) | 29 | 29 | 29 | 27 | 28 | 30
  Day 182 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [87.2 to 100] | 100 [87.7 to 100] | 100 [88.4 to 100]
  Day 385: number analyzed (Participants) | 0 | 0 | 29 | 27 | 0 | 0
  Day 385 |  |  | 100 [88.1 to 100] | 100 [87.2 to 100] |  |

2. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentrations - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Geometric mean concentrations (GMCs) were expressed in Elisa Unit per milliliter (EU/mL)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30
EU/mL
  Day 0: number analyzed (Participants) | 27 | 25 | 29 | 27 | 30 | 30
  Day 0 | 6935.6 [4974.4 to 9670.0] | 6841.5 [4954.4 to 9447.5] | 14381.9 [10313.7 to 20054.7] | 14552.3 [10670.0 to 19847.2] | 12799.7 [10297.3 to 15910.2] | 10888.1 [8004.1 to 14811.3]
  Day 21: number analyzed (Participants) | 28 | 25 | 29 | 27 | 30 | 30
  Day 21 | 45098.3 [34775.1 to 58486.2] | 37969.9 [26930.8 to 53534.1] | 46013.8 [33592.9 to 63027.5] | 27845.9 [20269.3 to 38254.5] | 25189.3 [20983.6 to 30238.0] | 16592.8 [13332.5 to 20650.4]
  Day 42: number analyzed (Participants) | 27 | 27 | 29 | 27 | 30 | 30
  Day 42 | 46177.1 [37510.4 to 56846.2] | 38598.2 [27818.0 to 53555.9] | 68348.8 [53244.4 to 87738.1] | 31718.0 [23755.4 to 42349.5] | 31665.4 [27405.9 to 36587.0] | 19681.1 [16293.6 to 23772.7]
  Day 182: number analyzed (Participants) | 29 | 29 | 29 | 27 | 28 | 30
  Day 182 | 21782.4 [17803.2 to 26651.0] | 24705.6 [18369.2 to 33227.7] | 33610.2 [26464.5 to 42685.3] | 17401.9 [13330.1 to 22717.5] | 20570.2 [16717.6 to 25310.5] | 15471.1 [11913.9 to 20090.4]
  Day 385: number analyzed (Participants) | 0 | 0 | 29 | 27 | 0 | 0
  Day 385 |  |  | 25346.9 [20205.0 to 31797.3] | 15768.2 [11999.3 to 20720.9] |  |

3. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seronegative subjects = concentration < 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. Seropositive subjects = concentration ≥ 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 132 EU/mL at post-vaccination. For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At Day 21 (post-vaccination 1 compared to pre-vaccination), Day 42 (post-vaccination 2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 27 | 25 | 29 | 27 | 30 | 30
Percentage of subjects
  Day 21: number analyzed (Participants) | 27 | 23 | 29 | 27 | 30 | 30
  Day 21 | 63.0 [42.4 to 80.6] | 52.2 [30.6 to 73.2] | 34.5 [17.9 to 54.3] | 7.4 [0.9 to 24.3] | 10.0 [2.1 to 26.5] | 6.7 [0.8 to 22.1]
  Day 42: number analyzed (Participants) | 25 | 25 | 29 | 27 | 30 | 30
  Day 42 | 72.0 [50.6 to 87.9] | 60.0 [38.7 to 78.9] | 55.2 [35.7 to 73.6] | 18.5 [6.3 to 38.1] | 20.0 [7.7 to 38.6] | 3.3 [0.1 to 17.2]

4. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. seropositive subjects = concentration ≥ 66 EU/mL for anti-H1 stalk ELISA prior to vaccination 10-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 330 EU/mL at post-vaccination, For initially seropositive subjects, antibody concentration at post-vaccination ≥ 10-fold the pre-vaccination antibody concentration.
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 27 | 25 | 29 | 27 | 30 | 30
Percentage of subjects
  Day 21: number analyzed (Participants) | 27 | 23 | 29 | 27 | 30 | 30
  Day 21 | 29.6 [13.8 to 50.2] | 34.8 [16.4 to 57.3] | 6.9 [0.8 to 22.8] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.6]
  Day 42: number analyzed (Participants) | 25 | 25 | 29 | 27 | 30 | 30
  Day 42 | 36.0 [18.0 to 57.5] | 28.0 [12.1 to 49.4] | 20.7 [8.0 to 39.7] | 7.4 [0.9 to 24.3] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.6]

5. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMC over pre-vaccination GMC.
Time Frame: At Day 21 (post-vaccination1/ pre-vaccination), Day 42 (post-vaccination2/ pre-vaccination), Day 182 (post-vaccination2/ pre-vaccination) and Day 385(post-vaccination2/ pre-vaccination - for H5N1 cohorts only )
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 27 | 25 | 29 | 27 | 30 | 30
Ratio
  Day 21: number analyzed (Participants) | 27 | 23 | 29 | 27 | 30 | 30
  Day 21 | 6.5 [4.7 to 9.2] | 5.9 [3.6 to 9.6] | 3.2 [2.3 to 4.5] | 1.9 [1.4 to 2.7] | 2.0 [1.6 to 2.4] | 1.5 [1.3 to 1.8]
  Day 42: number analyzed (Participants) | 25 | 25 | 29 | 27 | 30 | 30
  Day 42 | 7.0 [5.0 to 9.7] | 5.6 [3.6 to 8.7] | 4.8 [3.5 to 6.4] | 2.2 [1.6 to 3.0] | 2.5 [2.1 to 3.0] | 1.8 [1.5 to 2.1]
  Day 182: number analyzed (Participants) | 27 | 25 | 29 | 27 | 28 | 30
  Day 182 | 3.2 [2.4 to 4.1] | 3.6 [2.4 to 5.3] | 2.3 [1.8 to 3.1] | 1.2 [1.0 to 1.5] | 1.6 [1.4 to 1.9] | 1.4 [1.2 to 1.6]
  Day 385: number analyzed (Participants) | 0 | 0 | 29 | 27 | 0 | 0
  Day 385 |  |  | 1.8 [1.4 to 2.2] | 1.1 [0.9 to 1.3] |  |

6. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Equal or Above the Cut-off of 66 EU/mL - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with concentrations greater or equal than 66 Elisa Unit per milliliter (EU/mL)
Time Frame: At Day 0 (Pre-vaccination), Day 21 (Post-vaccination 1), Day 42 (Post-vaccination 2) and Day 385 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS | H5N1_PCN
Number analyzed (Participants) | 33 | 19
Percentage of subjects
  Day 0: number analyzed (Participants) | 32 | 17
  Day 0 | 100 [89.1 to 100] | 100 [80.5 to 100]
  Day 21: number analyzed (Participants) | 33 | 18
  Day 21 | 100 [89.4 to 100] | 100 [81.5 to 100]
  Day 42: number analyzed (Participants) | 33 | 18
  Day 42 | 100 [89.4 to 100] | 100 [81.5 to 100]
  Day 385: number analyzed (Participants) | 24 | 19
  Day 385 | 100 [85.8 to 100] | 100 [82.4 to 100]

7. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentrations -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 2
Time Frame: At Day 0 (Pre-vaccination), Day 21 (Post-vaccination 1), Day 42 (Post-vaccination 2) and Day 385 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_PAS | H5N1_PCN
Number analyzed (Participants) | 33 | 19
EU/mL
  Day 0: number analyzed (Participants) | 32 | 17
  Day 0 | 2075.4 [1458.3 to 2953.6] | 2123.2 [1042.1 to 4325.7]
  Day 21: number analyzed (Participants) | 33 | 18
  Day 21 | 16552.4 [9239.4 to 29653.7] | 2203.3 [1237.8 to 3922.1]
  Day 42: number analyzed (Participants) | 33 | 18
  Day 42 | 22195.2 [14601.3 to 33738.6] | 2272.1 [1310.1 to 3940.6]
  Day 385: number analyzed (Participants) | 24 | 19
  Day 385 | 8661.1 [5352.5 to 14014.8] | 2394.7 [1446.6 to 3964.0]

8. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 3
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS | H5N1_PCN
Number analyzed (Participants) | 32 | 17
Percentage of subjects
  Day 21 | 59.4 [40.6 to 76.3] | 0.0 [0.0 to 19.5]
  Day 42: number analyzed (Participants) | 32 | 16
  Day 42 | 71.9 [53.3 to 86.3] | 0.0 [0.0 to 20.6]

9. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 4
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS | H5N1_PCN
Number analyzed (Participants) | 32 | 17
Percentage of subjects
  Day 21 | 40.6 [23.7 to 59.4] | 0.0 [0.0 to 19.5]
  Day 42: number analyzed (Participants) | 32 | 16
  Day 42 | 53.1 [34.7 to 70.9] | 0.0 [0.0 to 20.6]

10. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 5
Time Frame: At Day 21 (post-vaccination1/ pre-vaccination), Day 42 (post-vaccination2/ pre-vaccination) and Day 385(post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS | H5N1_PCN
Number analyzed (Participants) | 32 | 17
Ratio
  Day 21 | 8.8 [5.0 to 15.6] | 1.1 [0.9 to 1.2]
  Day 42: number analyzed (Participants) | 32 | 16
  Day 42 | 11.3 [7.3 to 17.7] | 1.0 [0.8 to 1.2]
  Day 385: number analyzed (Participants) | 23 | 16
  Day 385 | 4.1 [2.3 to 7.2] | 1.4 [1.0 to 2.2]

11. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Equal or Above the Cut-off of 66 EU/mL - Adult Q-PAN-005 Cohort
Description: as for outcome 6
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 1), Day 182 (post-vaccination 1), Day 224 (Post-vaccination 2), Day 549 (post-vaccination 2), Day 591 (Post-vaccination 3) and Day 729 (Post-vaccination 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0 | 100 [86.8 to 100] | 100 [88.1 to 100]
  Day 42: number analyzed (Participants) | 26 | 28
  Day 42 | 100 [86.8 to 100] | 100 [87.7 to 100]
  Day 182 | 100 [86.8 to 100] | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 26 | 28
  Day 224 | 100 [86.8 to 100] | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 100 [85.8 to 100] | 100 [83.2 to 100]

12. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentrations - Adult Q-PAN-005 Cohort
Description: as for outcome 2
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
EU/mL
  Day 0 | 8946.2 [6147.1 to 13019.9] | 9205.1 [6434.5 to 13168.6]
  Day 42: number analyzed (Participants) | 26 | 28
  Day 42 | 35325.3 [25353.6 to 49218.9] | 10171.2 [7035.3 to 14705.0]
  Day 182 | 22057.9 [15456.7 to 31478.3] | 10123.1 [6701.6 to 15291.4]
  Day 224: number analyzed (Participants) | 26 | 28
  Day 224 | 18748.2 [13219.8 to 26588.7] | 43267.9 [31807.8 to 58856.9]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 21272.5 [16188.8 to 27952.7] | 23507.6 [16503.6 to 33484.1]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 29023.7 [22329.1 to 37725.4] | 33113.7 [23879.1 to 45919.6]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 22445.9 [17120.0 to 29428.7] | 21894.3 [15168.5 to 31602.4]

13. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. seropositive subjects = concentration ≥ 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 132 EU/mL at post-vaccination. For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: For group C: At Day 42 (post-dose1 compared to [/]Day 0), Day 224 (post-dose 2/Day 0), Day 591 (post-dose3 / Day 0) - For group G: At Day 224 (post-dose2 / Day 182); at Day 591 (post-dose3 / Day 182)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 50.0 [29.9 to 70.1] |
  Day 224 | 15.4 [4.4 to 34.9] | 46.4 [27.5 to 66.1]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 29.2 [12.6 to 51.1] | 50.0 [27.2 to 72.8]

14. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all subjects in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. seropositive subjects = concentration ≥ 66 EU/mL for anti-H1 stalk ELISA prior to vaccination 10-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 330 EU/mL at post-vaccination, For initially seropositive subjects, antibody concentration at post-vaccination ≥ 10-fold the pre-vaccination antibody concentration. The ≥10-fold increases were only calculated relative to baseline.
Time Frame: For group C: At Day 42 (post-dose1 compared to [/]Day 0), Day 224 (post-dose 2/Day 0), Day 591 (post-dose3 / Day 0) - For group G: At Day 224 (post-dose2 / Day 182), at Day 591 (post-dose3 / Day 182)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 23.1 [9.0 to 43.6] |
  Day 224 | 0.0 [0.0 to 13.2] | 25.0 [10.7 to 44.9]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 4.2 [0.1 to 21.1] | 5.0 [0.1 to 24.9]

15. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 5
Time Frame: At Day[D] 42 (post-dose[ps-d]1), D182 (ps-d1), D224 (ps-d2), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D0 for Group C and at D224 (ps-d2), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D182 for Group G
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 3.9 [2.8 to 5.6] |
  Day 182: number analyzed (Participants) | 26 | 0
  Day 182 | 2.5 [2.0 to 3.1] |
  Day 224 | 2.1 [1.7 to 2.6] | 4.0 [2.5 to 6.4]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 2.3 [1.7 to 3.1] | 2.0 [1.5 to 2.8]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 3.1 [2.2 to 4.2] | 2.9 [1.9 to 4.3]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 2.4 [1.8 to 3.2] | 1.9 [1.3 to 2.7]

16. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Equal or Above the Cut-off of 66 EU/mL - Adult H5N1-012 Cohort
Description: as for outcome 6
Time Frame: At D0 (Pre), D21 (Post-dose 1), Month (M)6 (post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Day 21 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 100 [93.0 to 100] | 100 [92.7 to 100]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 100 [92.9 to 100] | 100 [92.6 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 100 [92.6 to 100] | 100 [92.5 to 100]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 100 [92.7 to 100] | 100 [92.1 to 100]

17. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentrations - Adult H5N1-012 Cohort
Description: as for outcome 2
Time Frame: At D0 (Pre), D21 (Post-dose 1), Month (M)6 (post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
EU/mL
  Day 0 | 9340.1 [7411.6 to 11770.5] | 8409.3 [6746.1 to 10482.4]
  Day 21 | 35805.4 [29821.1 to 42990.6] | 40245.6 [31912.9 to 50753.9]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 16123.6 [13232.7 to 19646.1] | 17337.3 [13536.2 to 22206.0]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 14548.7 [11989.4 to 17654.2] | 16242.1 [12854.0 to 20523.3]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 32675.5 [27585.4 to 38704.8] | 37096.0 [29342.0 to 46899.1]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 21154.6 [17597.8 to 25430.2] | 19508.2 [15715.0 to 24217.0]

18. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult H5N1-012 Cohort
Description: as for outcome 13
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 39.6 [26.5 to 54.0] | 55.1 [40.2 to 69.3]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 39.6 [25.8 to 54.7] | 46.8 [32.1 to 61.9]

19. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult H5N1-012 Cohort
Description: as for outcome 14
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 15.1 [6.7 to 27.6] | 18.4 [8.8 to 32.0]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 14.6 [6.1 to 27.8] | 21.3 [10.7 to 35.7]

20. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult H5N1-012 Cohort
Description: as for outcome 5
Time Frame: At D21 (post-dose[ps-d]1), M6 (ps-d1), M12 (ps-d1), M12+21days (ps-d2) and M18 compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Ratio
  Day 21 | 3.8 [3.0 to 5.0] | 4.8 [3.7 to 6.2]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 1.7 [1.5 to 2.1] | 2.1 [1.7 to 2.5]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.6 [1.4 to 1.8] | 1.9 [1.6 to 2.4]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 3.6 [2.8 to 4.8] | 4.5 [3.4 to 6.0]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 2.3 [1.8 to 2.9] | 2.5 [1.9 to 3.1]

21. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentration Equal or Above the Cut-off of 66 EU/mL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 6
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 100 [88.4 to 100]
  Day 21 | 100 [88.4 to 100]

22. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Concentrations - Adult FLU D-QIV-015 Cohort
Description: as for outcome 2
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
EU/mL
  Day 0 | 11215.8 [8015.8 to 15693.3]
  Day 21 | 30437.5 [24261.2 to 38186.2]

23. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult FLU D-QIV-015 Cohort
Description: as for outcome 3
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 33.3 [17.3 to 52.8]

24. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk ELISA Antibody Concentration - Adult FLU D-QIV-015 Cohort
Description: as for outcome 4
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 3.3 [0.1 to 17.2]

25. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult FLU D-QIV-015 Cohort
Description: as for outcome 5
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Ratio | 2.7 [2.0 to 3.7]

26. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by microneutralization (MN) for all subjects who received an adjuvant system (AS) vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/Dilution (1/DIL).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 0 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 21 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 42 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 182: number analyzed (Participants) | 29 | 29 | 28
  Day 182 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [87.7 to 100]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 100 [88.1 to 100] |

27. Primary Outcome: Anti-H1 Stalk Antibody Titers (by MN) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, Geometric mean titers (GMTs) were calculated with 95% CI for each treatment group within each study cohort.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Titer
  Day 0 | 11.0 [10.0 to 12.1] | 18.6 [14.4 to 24.1] | 30.3 [19.1 to 48.2]
  Day 21 | 30.8 [23.1 to 40.9] | 40.0 [29.0 to 55.2] | 60.6 [37.9 to 96.9]
  Day 42 | 33.0 [25.7 to 42.6] | 64.5 [47.0 to 88.5] | 91.9 [62.0 to 136.1]
  Day 182: number analyzed (Participants) | 29 | 29 | 28
  Day 182 | 18.2 [14.3 to 23.1] | 44.0 [31.9 to 60.7] | 58.0 [35.4 to 95.0]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 33.0 [25.2 to 43.4] |

28. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for anti-H1 stalk MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for anti-H1 stalk MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 21 | 44.8 [26.4 to 64.3] | 27.6 [12.7 to 47.2] | 23.3 [9.9 to 42.3]
  Day 42 | 51.7 [32.5 to 70.6] | 65.5 [45.7 to 82.1] | 46.7 [28.3 to 65.7]

29. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk Antibody Titer (by MN) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for anti-H1 stalk MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for anti-H1 stalk MN prior to vaccination. 10-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 50 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 10-fold the pre-vaccination antibody titer.
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 21 | 6.9 [0.8 to 22.8] | 6.9 [0.8 to 22.8] | 6.7 [0.8 to 22.1]
  Day 42 | 6.9 [0.8 to 22.8] | 6.9 [0.8 to 22.8] | 6.7 [0.8 to 22.1]

30. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMT over pre-vaccination GMT.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Ratio
  Day 21 | 2.8 [2.0 to 3.8] | 2.1 [1.6 to 2.9] | 2.0 [1.4 to 2.8]
  Day 42 | 3.0 [2.3 to 4.0] | 3.5 [2.6 to 4.6] | 3.0 [2.2 to 4.1]
  Day 182: number analyzed (Participants) | 29 | 29 | 28
  Day 182 | 1.7 [1.3 to 2.1] | 2.4 [1.7 to 3.3] | 2.0 [1.4 to 2.8]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 1.8 [1.3 to 2.4] |

31. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titerss greater or equal than 10 1/DIL.
Time Frame: At Day 0 (Pre-vaccination), Day 21 (Post-vaccination 1), Day 42 (Post-vaccination 2) and Day 385 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 0 | 100 [89.4 to 100]
  Day 21 | 100 [89.4 to 100]
  Day 42 | 100 [89.4 to 100]
  Day 385: number analyzed (Participants) | 30
  Day 385 | 100 [89.4 to 100]

32. Primary Outcome: Anti-H1 Stalk Antibody Titers (by MN) -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 27
Time Frame: At Day 0 (Pre-vaccination), Day 21 (Post-vaccination 1), Day 42 (Post-vaccination 2) and Day 385 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Titer
  Day 0 | 19.2 [15.1 to 24.3]
  Day 21 | 43.5 [30.3 to 62.5]
  Day 42 | 44.4 [32.7 to 60.5]
  Day 385: number analyzed (Participants) | 30
  Day 385 | 22.4 [17.1 to 29.5]

33. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 28
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 21 | 39.4 [22.9 to 57.9]
  Day 42 | 39.4 [22.9 to 57.9]

34. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 29
Time Frame: At Day 21 (post-vaccination1 compared to pre-vaccination), Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 21 | 6.1 [0.7 to 20.2]
  Day 42 | 3.0 [0.1 to 15.8]

35. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines
Description: as for outcome 30
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Ratio
  Day 21 | 2.3 [1.6 to 3.3]
  Day 42 | 2.3 [1.6 to 3.3]
  Day 385: number analyzed (Participants) | 30
  Day 385 | 1.1 [0.8 to 1.5]

36. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/DIL
Time Frame: Group C: At D0 (Pre), D42 (Post-dose 1), D182 (post-dose 1), D549 (post-dose 2), D591 (Post-dose 3) and D729 (Post-dose 3); Group G: At D182 (Post-dose 1), D224 (Post-dose 2), D549 (post-dose 2), D591 (Post-dose 3) and D729 (Post-dose 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 100 [86.8 to 100] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 100 [86.8 to 100] |
  Day 182 | 100 [86.8 to 100] | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 100 [85.8 to 100] | 100 [83.2 to 100]

37. Primary Outcome: Anti-H1 Stalk Enzyme-linked Immunosorbent Assay (ELISA) Antibody Titers - Adult Q-PAN-005 Cohort
Description: as for outcome 27
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Titer
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 18.5 [15.4 to 22.2] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 48.2 [34.9 to 66.5] |
  Day 182 | 40.0 [32.0 to 50.0] | 15.4 [13.3 to 17.8]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 51.2 [37.2 to 70.6]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 31.2 [23.4 to 41.4] | 27.8 [21.1 to 36.6]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 40.0 [31.8 to 50.3] | 40.0 [28.7 to 55.8]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 49.0 [38.7 to 62.0] | 36.1 [26.6 to 48.8]

38. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for anti-H1 stalk MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for anti-H1 stalk MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: For group C: At Day 42 (post-dose1 compared to [/]Day 0), at Day 591 (post-dose3 / Day 0) - For group G: At Day 224 (post-dose2 / Day 182), at Day 591 (post-dose3 / Day 182)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 42.3 [23.4 to 63.1] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 57.1 [37.2 to 75.5]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 25.0 [9.8 to 46.7] | 45.0 [23.1 to 68.5]

39. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for anti-H1 stalk MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for anti-H1 stalk MN prior to vaccination. 10-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 50 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 10-fold the pre-vaccination antibody titer. The ≥10-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 7.7 [0.9 to 25.1] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 7.1 [0.9 to 23.5]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 16.8]

40. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 30
Time Frame: At Day[D] 42 (post-dose[ps-d]1), D182 (ps-d1), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D0 for Group C and at D224 (ps-d2), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D182 for Group G
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 2.6 [1.8 to 3.9] |
  Day 182: number analyzed (Participants) | 26 | 0
  Day 182 | 2.2 [1.7 to 2.8] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 3.3 [2.4 to 4.5]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 1.7 [1.2 to 2.4] | 1.8 [1.3 to 2.3]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 2.1 [1.6 to 2.8] | 2.5 [1.8 to 3.6]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 2.6 [1.9 to 3.5] | 2.3 [1.7 to 3.1]

41. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult H5N1-012 Cohort
Description: as for outcome 36
Time Frame: At D0 (Pre), D21 (Post-dose 1), Month (M)6 (post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Day 21 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 100 [93.0 to 100] | 100 [92.7 to 100]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 100 [92.9 to 100] | 100 [92.6 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 100 [92.6 to 100] | 100 [92.5 to 100]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 100 [92.7 to 100] | 97.8 [88.2 to 99.9]

42. Primary Outcome: Anti-H1 Stalk Antibody Titers (by MN) - Adult H5N1-012 Cohort
Description: as for outcome 27
Time Frame: At D0 (Pre), D21 (Post-dose 1), Month (M)6 (post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Titer
  Day 0 | 19.0 [15.8 to 22.8] | 26.5 [21.9 to 32.1]
  Day 21 | 56.9 [45.8 to 70.8] | 106.2 [84.1 to 134.0]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 30.1 [25.6 to 35.3] | 29.3 [24.1 to 35.6]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 25.3 [21.6 to 29.6] | 40.6 [32.6 to 50.5]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 40.0 [33.1 to 48.4] | 74.3 [59.1 to 93.5]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 32.4 [27.1 to 38.7] | 32.7 [26.5 to 40.4]

43. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Adult H5N1-012 Cohort
Description: as for outcome 38
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 49.1 [35.1 to 63.2] | 67.3 [52.5 to 80.1]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 31.3 [18.7 to 46.3] | 51.1 [36.1 to 65.9]

44. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk Antibody Titer - Adult H5N1-012 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H1 stalk antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for anti-H1 stalk MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for anti-H1 stalk MN prior to vaccination. 10-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 50 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 10-fold the pre-vaccination antibody titer. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 9.4 [3.1 to 20.7] | 12.2 [4.6 to 24.8]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 4.2 [0.5 to 14.3] | 6.4 [1.3 to 17.5]

45. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult H5N1-012 Cohort
Description: as for outcome 30
Time Frame: At D21 (post-dose[ps-d]1), M6 (ps-d1), M12 (ps-d1), M12+21days (ps-d2) and M18 compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Ratio
  Day 21 | 3.0 [2.3 to 3.9] | 4.0 [3.1 to 5.1]
  Month 6: number analyzed (Participants) | 51 | 49
  Month 6 | 1.6 [1.3 to 2.0] | 1.1 [0.9 to 1.4]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.3 [1.1 to 1.6] | 1.5 [1.2 to 1.9]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 2.1 [1.6 to 2.7] | 2.9 [2.2 to 3.8]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 1.7 [1.4 to 2.2] | 1.3 [1.0 to 1.7]

46. Primary Outcome: Percentage of Subjects With Anti-H1 Stalk Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 36
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 100 [88.4 to 100]
  Day 21 | 100 [88.4 to 100]

47. Primary Outcome: Anti-H1 Stalk Antibody Titers (by MN) - Adult FLU D-QIV-015 Cohort
Description: as for outcome 27
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Titer
  Day 0 | 28.3 [22.9 to 35.0]
  Day 21 | 76.4 [57.3 to 101.9]

48. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H1 Stalk Antibody Titer by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 28
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 53.3 [34.3 to 71.7]

49. Primary Outcome: Percentage of Subjects With a ≥10-fold Rise for Anti-H1 Stalk Antibody Titer - Adult FLU D-QIV-015 Cohort
Description: as for outcome 29
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 10.0 [2.1 to 26.5]

50. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 30
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Ratio | 2.7 [1.8 to 4.0]

51. Primary Outcome: Percentage of Subjects With Anti-H2 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with concentrations greater or equal than 50 Elisa Unit per milliliter (EU/mL)
Time Frame: At Day 42 (Post-vaccination 2), and final timepoint (for persistence) (i.e., Day 182 for the Q-Pan-H1N1-019, Q-PAN-H9N2-001 and Day 385 for the CC-Pan-H5N1 study cohorts)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 0: number analyzed (Participants) | 27 | 29 | 30
  Day 0 | 100 [87.2 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 42: number analyzed (Participants) | 27 | 29 | 30
  Day 42 | 100 [87.2 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 182: number analyzed (Participants) | 29 | 0 | 28
  Day 182 | 100 [88.1 to 100] |  | 100 [87.7 to 100]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 100 [88.1 to 100] |

52. Primary Outcome: Anti-H2 Full Length HA ELISA Antibody Concentrations - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Geometric mean concentrations (GMCs) were expressed in Elisa Unit per milliliter (EU/mL)
Time Frame: as for outcome 51
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
EU/mL
  Day 0: number analyzed (Participants) | 27 | 29 | 30
  Day 0 | 3697.2 [2695.5 to 5071.1] | 8366.5 [5770.6 to 12130.2] | 14704.5 [10160.7 to 21280.2]
  Day 42: number analyzed (Participants) | 27 | 29 | 30
  Day 42 | 20783.2 [16291.5 to 26513.4] | 51118.1 [39968.6 to 65378.0] | 36716.0 [27343.3 to 49301.5]
  Day 182: number analyzed (Participants) | 29 | 0 | 28
  Day 182 | 12674.3 [9909.2 to 16210.9] |  | 23927.1 [17505.5 to 32704.2]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 19903.0 [15283.4 to 25919.0] |

53. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H2 Full Length HA ELISA Antibody Concentration - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 25 | 29 | 30
Percentage of subjects | 72.0 [50.6 to 87.9] | 62.1 [42.3 to 79.3] | 20.0 [7.7 to 38.6]

54. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H2 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMC over pre-vaccination GMC.
Time Frame: At Day 42 (post-vaccination2/ Day 0), and final timepoint (for persistence) compared to Day 0 (i.e., Day 182 for the Q-Pan-H1N1-019, Q-PAN-H9N2-001 and Day 385 for the CC-Pan-H5N1 study cohorts)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 25 | 29 | 30
Ratio
  Day 42 | 6.0 [4.4 to 8.0] | 6.1 [4.3 to 8.7] | 2.5 [2.0 to 3.1]
  Day 182: number analyzed (Participants) | 25 | 0 | 28
  Day 182 | 3.5 [2.8 to 4.4] |  | 1.8 [1.5 to 2.1]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 2.4 [1.9 to 3.0] |

55. Primary Outcome: Percentage of Subjects With Anti-H2 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 51
Time Frame: At Day 42 (Post-vaccination 2) and final timepoint (for persistence) (i.e., Day 385)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 42 | 100 [89.4 to 100]
  Day 385: number analyzed (Participants) | 24
  Day 385 | 100 [85.8 to 100]

56. Primary Outcome: Anti-H2 Full Length HA ELISA Antibody Concentrations -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 52
Time Frame: At Day 42 (Post-vaccination 2) and final timepoint (for persistence) (i.e., Day 385)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
EU/mL
  Day 42 | 20542.9 [15121.2 to 27908.4]
  Day 385: number analyzed (Participants) | 24
  Day 385 | 7258.3 [4703.9 to 11199.9]

57. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H2 Full Length HA ELISA Antibody Concentration - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohortand for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At Day 42 (post-vaccination2 compared to Day 0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 29
Percentage of subjects | 96.6 [82.2 to 99.9]

58. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H2 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 54
Time Frame: At Day 42 (post-vaccination2/ Day 0) and final time point (for persistence)(i.e., Day 385[post-vaccination2]/ Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 29
Ratio
  Day 42 | 17.1 [11.7 to 25.1]
  Day 385: number analyzed (Participants) | 22
  Day 385 | 5.5 [3.1 to 9.8]

59. Primary Outcome: Percentage of Subjects With Anti-H2 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult Q-PAN-005 Cohort
Description: as for outcome 51
Time Frame: At D0(Pre), D42(Post-dose [Pst-d]1), D182(Pst-d1), D549(Pst-d2), D591(Pst-d3) and D729(Pst-d3) for group C, and D182(Pst-d1), D224(Pst-d2), D549(Pst-d2), D591(Pst-d3) and D729(Pst-d3) for group G
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 100 [86.8 to 100] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 100 [86.8 to 100] |
  Day 182 | 100 [86.8 to 100] | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 100 [85.8 to 100] | 100 [83.2 to 100]

60. Primary Outcome: Anti-H2 Full Length HA ELISA Antibody Concentrations - Adult Q-PAN-005 Cohort
Description: as for outcome 52
Time Frame: as for outcome 59
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
EU/mL
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 5832.4 [4271.3 to 7964.0] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 23187.8 [16597.1 to 32395.7] |
  Day 182 | 15364.4 [11057.9 to 21347.9] | 6914.7 [4722.5 to 10124.4]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 34071.6 [25325.9 to 45837.3]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 12974.0 [10089.8 to 16682.7] | 15142.3 [10406.0 to 22034.2]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 21467.9 [16930.0 to 27222.1] | 24791.3 [18324.3 to 33540.7]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 14534.4 [11280.4 to 18727.3] | 13865.1 [9476.2 to 20286.9]

61. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H2 Full Length HA ELISA Antibody Concentration - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H2 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H2 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 50.0 [29.9 to 70.1] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 46.4 [27.5 to 66.1]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 45.8 [25.6 to 67.2] | 55.0 [31.5 to 76.9]

62. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H2 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 54
Time Frame: At Day[D] 42 (post-dose[ps-d]1), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D0 for Group C and at D224 (ps-d2), D549 (ps-d2), D591 (ps-d3) and D729(ps-d3) compared to D182 for Group G
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 4.0 [2.8 to 5.7] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 4.7 [3.0 to 7.3]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 2.2 [1.6 to 2.9] | 2.0 [1.5 to 2.6]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 3.6 [2.7 to 4.6] | 3.3 [2.2 to 4.8]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 4.7 [3.0 to 7.3] | 1.8 [1.3 to 2.5]

63. Primary Outcome: Percentage of Subjects With Anti-H2 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult H5N1-012 Cohort
Description: as for outcome 51
Time Frame: At D0 (Pre), D21 (Post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Day 21 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 100 [92.9 to 100] | 100 [92.6 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 100 [92.6 to 100] | 100 [92.5 to 100]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 100 [92.7 to 100] | 100 [92.1 to 100]

64. Primary Outcome: Anti-H2 Full Length HA ELISA Antibody Concentrations - Adult H5N1-012 Cohort
Description: as for outcome 52
Time Frame: At D0 (Pre), D21 (Post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
EU/mL
  Day 0 | 8735.3 [6375.6 to 11968.5] | 8633.4 [6344.7 to 11747.7]
  Day 21 | 34355.8 [26840.9 to 43974.8] | 40833.0 [31899.1 to 52269.0]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 14575.6 [11067.3 to 19196.0] | 15958.9 [12427.1 to 20494.4]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 48534.4 [39207.4 to 60080.4] | 51228.3 [40614.9 to 64615.3]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 23376.4 [18227.7 to 29979.3] | 20685.0 [16219.1 to 26380.5]

65. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H2 Full Length HA ELISA Antibody Concentration - Adult H5N1-012 Cohort
Description: as for outcome 61
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 41.5 [28.1 to 55.9] | 51.0 [36.3 to 65.6]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 56.3 [41.2 to 70.5] | 61.7 [46.4 to 75.5]

66. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H2 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult H5N1-012 Cohort
Description: as for outcome 54
Time Frame: At D21 (post-dose[ps-d]1), M12 (ps-d1), M12+21days (ps-d2) and M18 compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Ratio
  Day 21 | 3.9 [3.0 to 5.1] | 4.7 [3.7 to 6.1]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.7 [1.4 to 2.0] | 1.8 [1.5 to 2.3]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 5.6 [4.0 to 8.0] | 6.1 [4.5 to 8.1]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 2.6 [1.9 to 3.6] | 2.5 [2.0 to 3.2]

67. Primary Outcome: Percentage of Subjects With Anti-H2 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 51
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 100 [88.4 to 100]
  Day 21 | 100 [88.4 to 100]

68. Primary Outcome: Anti-H2 Full Length HA ELISA Antibody Concentrations - Adult FLU D-QIV-015 Cohort
Description: as for outcome 52
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
EU/mL
  Day 0 | 6435.6 [4852.3 to 8535.5]
  Day 21 | 12074.6 [9400.2 to 15509.9]

69. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H2 Full Length HA ELISA Antibody Concentration - Adult FLU D-QIV-015 Cohort
Description: as for outcome 53
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 6.7 [0.8 to 22.1]

70. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H2 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult FLU D-QIV-015 Cohort
Description: as for outcome 54
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Ratio | 1.9 [1.6 to 2.2]

71. Primary Outcome: Percentage of Subjects With Anti-H18 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with concentrations greater or equal than 50 Elisa Unit per milliliter (EU/mL)
Time Frame: as for outcome 51
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 42: number analyzed (Participants) | 27 | 29 | 30
  Day 42 | 100 [87.2 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 182: number analyzed (Participants) | 29 | 0 | 28
  Day 182 | 100 [88.1 to 100] |  | 100 [87.7 to 100]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 100 [88.1 to 100] |

72. Primary Outcome: Anti-H18 Full Length HA ELISA Antibody Concentrations - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Geometric mean concentrations (GMCs) were expressed in Elisa Unit per milliliter (EU/mL)
Time Frame: as for outcome 51
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
EU/mL
  Day 42: number analyzed (Participants) | 27 | 29 | 30
  Day 42 | 15959.9 [12897.9 to 19748.9] | 28492.2 [21814.5 to 37214.0] | 19636.8 [16519.2 to 23342.8]
  Day 182: number analyzed (Participants) | 29 | 0 | 28
  Day 182 | 7791.5 [6301.3 to 9634.2] |  | 9859.5 [7806.5 to 12452.5]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 11491.9 [8848.8 to 14924.5] |

73. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H18 Full Length HA ELISA Antibody Concentration - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 25 | 29 | 30
Percentage of subjects | 48.0 [27.8 to 68.7] | 51.7 [32.5 to 70.6] | 30.0 [14.7 to 49.4]

74. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H18 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMC over pre-vaccination GMC.
Time Frame: as for outcome 54
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 27 | 29 | 30
Ratio
  Day 42: number analyzed (Participants) | 25 | 29 | 30
  Day 42 | 5.3 [3.6 to 8.0] | 4.9 [3.5 to 6.9] | 2.8 [2.3 to 3.5]
  Day 182: number analyzed (Participants) | 27 | 0 | 28
  Day 182 | 2.5 [1.8 to 3.4] |  | 1.4 [1.2 to 1.8]
  Day 385: number analyzed (Participants) | 0 | 29 | 0
  Day 385 |  | 2.0 [1.6 to 2.5] |

75. Primary Outcome: Percentage of Subjects With Anti-H18 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 71
Time Frame: At Day 42 (Post-vaccination 2) and final timepoint (for persistence) (i.e., Day 385)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 42 | 100 [89.4 to 100]
  Day 385: number analyzed (Participants) | 24
  Day 385 | 100 [85.8 to 100]

76. Primary Outcome: Anti-H18 Full Length HA ELISA Antibody Concentrations -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 72
Time Frame: At Day 42 (Post-vaccination 2) and final timepoint (for persistence) (i.e., Day 385)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
EU/mL
  Day 42 | 12214.4 [8399.6 to 17761.9]
  Day 385: number analyzed (Participants) | 24
  Day 385 | 3974.2 [2548.8 to 6196.8]

77. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H18 Full Length HA ELISA Antibody Concentration - Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohortand for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At Day 42 (post-vaccination2 compared to Day 0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects | 81.8 [64.5 to 93.0]

78. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H18 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination -Pediatric Q-PAN H5N1-AS03-021 Cohort
Description: as for outcome 74
Time Frame: At Day 42 (post-vaccination2/ Day 0) and final time point (for persistence)(i.e., Day 385(post-vaccination2/ Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Ratio
  Day 42 | 15.9 [9.9 to 25.6]
  Day 385: number analyzed (Participants) | 24
  Day 385 | 4.7 [2.7 to 8.4]

79. Primary Outcome: Percentage of Subjects With Anti-H18 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult Q-PAN-005 Cohort
Description: as for outcome 71
Time Frame: At D0(Pre), D42 (Post-dose[Pst-d]1), D182(Pst-d1), D549(Pst-d2), D591(Pst-d3) and D729(Pst-d3) for group C, and D182(Pst-d1), D224(Pst-d2), D549(Pst-d2), D591(Pst-d3) and D729(Pst-d3) for group G
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 100 [86.8 to 100] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 100 [86.8 to 100] |
  Day 182 | 100 [86.8 to 100] | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 100 [85.8 to 100] | 100 [83.2 to 100]

80. Primary Outcome: Anti-H18 Full Length HA ELISA Antibody Concentrations - Adult Q-PAN-005 Cohort
Description: as for outcome 72
Time Frame: as for outcome 79
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
EU/mL
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 4858.6 [3288.8 to 7177.6] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 21291.6 [15138.2 to 29946.1] |
  Day 182 | 10859.0 [7483.4 to 15757.2] | 4268.3 [2736.3 to 6658.1]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 20162.7 [14733.6 to 27592.3]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 10935.8 [8226.0 to 14538.4] | 12308.9 [8353.2 to 18138.0]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 15362.8 [11801.3 to 19999.2] | 14064.2 [9991.3 to 19797.4]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 11917.5 [8775.7 to 16184.0] | 10921.9 [7313.7 to 16310.4]

81. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H18 Full Length HA ELISA Antibody Concentration - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of anti-H18 antibody by ELISA for the subjects who received an AS vaccine in each study cohort and for the subjects in the FLU D-QIV-015 study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = concentration < 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. seropositive subjects = concentration ≥ 50 EU/mL for anti-H18 HA (full length) antibody prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 100 EU/mL at post-vaccination; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 46.2 [26.6 to 66.6] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 46.4 [27.5 to 66.1]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 37.5 [18.8 to 59.4] | 40.0 [19.1 to 63.9]

82. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H18 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 74
Time Frame: as for outcome 62
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 4.4 [3.1 to 6.3] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 4.5 [2.7 to 7.3]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 2.2 [1.6 to 2.9] | 2.5 [1.7 to 3.5]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 3.0 [2.1 to 4.2] | 2.8 [1.9 to 4.2]
  Day 729: number analyzed (Participants) | 24 | 20
  Day 729 | 2.3 [1.7 to 3.2] | 2.2 [1.6 to 3.1]

83. Primary Outcome: Percentage of Subjects With Anti-H18 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult H5N1-012 Cohort
Description: as for outcome 71
Time Frame: At D0 (Pre), D21 (Post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Day 21 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 100 [92.9 to 100] | 100 [92.6 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 100 [92.6 to 100] | 100 [92.5 to 100]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 100 [92.7 to 100] | 100 [92.1 to 100]

84. Primary Outcome: Anti-H18 Full Length HA ELISA Antibody Concentrations - Adult H5N1-012 Cohort
Description: as for outcome 72
Time Frame: At D0 (Pre), D21 (Post-dose 1), M12 (Post-dose1), M12+21days (post-dose2), M18 (Post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
EU/mL
  Day 0 | 5105.9 [3937.3 to 6621.4] | 4856.6 [3949.9 to 5971.6]
  Day 21 | 22141.6 [18114.4 to 27064.1] | 21054.9 [16966.2 to 26129.0]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 6743.4 [5489.0 to 8284.6] | 7249.2 [5785.2 to 9083.6]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 14532.2 [12132.7 to 17406.2] | 16655.6 [13122.9 to 21139.2]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 9467.3 [7750.0 to 11565.2] | 10315.9 [8230.5 to 12929.6]

85. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H18 Full Length HA ELISA Antibody Concentration - Adult H5N1-012 Cohort
Description: as for outcome 81
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 37.7 [24.8 to 52.1] | 46.9 [32.5 to 61.7]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 31.3 [18.7 to 46.3] | 34.0 [20.9 to 49.3]

86. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H18 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult H5N1-012 Cohort
Description: as for outcome 74
Time Frame: At D21 (post-dose[ps-d]1), M12 (ps-d1), M12+21days (ps-d2) and M18 compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Ratio
  Day 21 | 4.3 [3.2 to 5.8] | 4.3 [3.4 to 5.6]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.4 [1.2 to 1.6] | 1.5 [1.2 to 1.8]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 3.0 [2.3 to 4.1] | 3.5 [2.7 to 4.5]
  Month 18: number analyzed (Participants) | 49 | 45
  Month 18 | 1.9 [1.5 to 2.5] | 2.3 [1.8 to 2.9]

87. Primary Outcome: Percentage of Subjects With Anti-H18 Full Length HA ELISA Antibody Concentration Equal or Above the Cut-off of 50 EU/mL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 71
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 100 [88.4 to 100]
  Day 21 | 100 [88.4 to 100]

88. Primary Outcome: Anti-H18 Full Length HA ELISA Antibody Concentrations - Adult FLU D-QIV-015 Cohort
Description: as for outcome 72
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
EU/mL
  Day 0 | 5950.9 [4212.2 to 8407.4]
  Day 21 | 11025.1 [8572.8 to 14178.9]

89. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for Anti-H18 Full Length HA ELISA Antibody Concentration - Adult FLU D-QIV-015 Cohort
Description: as for outcome 73
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 13.3 [3.8 to 30.7]

90. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H18 Full Length HA ELISA Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult FLU D-QIV-015 Cohort
Description: as for outcome 74
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Ratio | 1.9 [1.4 to 2.4]

91. Primary Outcome: Percentage of Subjects With RG Reassortant Virus (H5N8) Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/Dilution )
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects
  Day 0 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]
  Day 42 | 100 [88.1 to 100] | 100 [88.1 to 100] | 100 [88.4 to 100]

92. Primary Outcome: RG Reassortant Virus (H5N8) Antibody Titers (by MN) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, Geometric mean titers (GMTs) were calculated with 95% CI for each treatment group within each study cohort.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Titer
  Day 0 | 14.3 [12.1 to 16.9] | 23.6 [16.9 to 33.1] | 30.3 [23.6 to 39.0]
  Day 42 | 46.2 [34.1 to 62.5] | 78.1 [54.0 to 113.0] | 72.9 [55.7 to 95.5]

93. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for RG Reassortant Virus (H5N8) Antibody Titer by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination. seropositive subjects = titer ≥ 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Percentage of subjects | 55.2 [35.7 to 73.6] | 51.7 [32.5 to 70.6] | 43.3 [25.5 to 62.6]

94. Primary Outcome: Mean Geometric Increase (MGI) for RG Reassortant Virus (H5N8) Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMT over pre-vaccination GMT.
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 29 | 29 | 30
Ratio | 3.2 [2.4 to 4.4] | 3.3 [2.5 to 4.5] | 2.4 [1.9 to 3.1]

95. Primary Outcome: Percentage of Subjects With RG Reassortant Virus (H5N8) Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titerss greater or equal than 10 1/DIL.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 0 | 97.0 [84.2 to 99.9]
  Day 42 | 100 [89.4 to 100]

96. Primary Outcome: RG Reassortant Virus (H5N8) Antibody Titers (by MN) -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 92
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Titer
  Day 0 | 14.3 [11.6 to 17.5]
  Day 42 | 48.3 [38.0 to 61.4]

97. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for RG Reassortant Virus (H5N8) Antibody Titer by MN - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects | 54.5 [36.4 to 71.9]

98. Primary Outcome: Mean Geometric Increase (MGI) for RG Reassortant Virus (H5N8) Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 94
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Ratio | 3.4 [2.5 to 4.5]

99. Primary Outcome: Percentage of Subjects With RG Reassortant Virus (H5N8) Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/DIL
Time Frame: Group C: At D0 (Pre), D42 (Post-dose 1), D549 (post-dose 2) and D591 (Post-dose 3); Group G: At D182 (Post-dose 1), D224 (Post-dose 2), D549 (post-dose 2) and D591 (Post-dose 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 100 [86.8 to 100] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 100 [86.8 to 100] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]

100. Primary Outcome: RG Reassortant Virus (H5N8) Enzyme-linked Immunosorbent Assay (ELISA) Antibody Titers - Adult Q-PAN-005 Cohort
Description: as for outcome 92
Time Frame: as for outcome 99
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Titer
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 20.0 [15.2 to 26.3] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 34.1 [26.8 to 43.4] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 19.5 [17.1 to 22.3]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 51.2 [36.3 to 72.3]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 27.1 [22.1 to 33.3] | 27.8 [22.5 to 34.5]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 155.4 [103.2 to 234.0] | 82.8 [58.9 to 116.4]

101. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for RG Reassortant Virus (H5N8) Antibody Titer by MN - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of RG reassortant virus (H5N8) antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination. seropositive subjects = titer ≥ 10 1/DIL for RG reassortant virus (H5N8) MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 26.9 [11.6 to 47.8] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 42.9 [24.5 to 62.8]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 83.3 [62.6 to 95.3] | 55.0 [31.5 to 76.9]

102. Primary Outcome: Mean Geometric Increase (MGI) for RG Reassortant Virus (H5N8) Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 94
Time Frame: At Day[D] 42 (post-dose[ps-d]1), D549 (ps-d2) and D591 (ps-d3) compared to D0 for Group C and at D224 (ps-d2), D549 (ps-d2) and D591 (ps-d3) compared to D182 for Group G
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 1.7 [1.1 to 2.5] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 2.6 [1.9 to 3.7]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 1.4 [1.0 to 1.8] | 1.3 [1.0 to 1.7]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 7.8 [4.7 to 12.9] | 4.0 [2.7 to 5.9]

103. Primary Outcome: Percentage of Subjects With RG Reassortant Virus (H5N8) Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult H5N1-012 Cohort
Description: as for outcome 99
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Day 21 | 100 [93.3 to 100] | 100 [92.7 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 100 [92.6 to 100] | 100 [92.5 to 100]

104. Primary Outcome: RG Reassortant Virus (H5N8) Antibody Titers (by MN) - Adult H5N1-012 Cohort
Description: as for outcome 92
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Titer
  Day 0 | 20.0 [17.2 to 23.2] | 18.9 [17.0 to 21.0]
  Day 21 | 40.5 [32.7 to 50.2] | 44.8 [36.4 to 55.2]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 146.7 [108.3 to 198.9] | 256.5 [181.6 to 362.2]

105. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for RG Reassortant Virus (H5N8) Antibody Titer by MN - Adult H5N1-012 Cohort
Description: as for outcome 101
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 21 | 34.0 [21.5 to 48.3] | 30.6 [18.3 to 45.4]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 77.1 [62.7 to 88.0] | 91.5 [79.6 to 97.6]

106. Primary Outcome: Mean Geometric Increase (MGI) for RG Reassortant Virus (H5N8) Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult H5N1-012 Cohort
Description: as for outcome 94
Time Frame: At D21 (post-dose[ps-d]1), M12 (ps-d1) and M12+21days (ps-d2) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Ratio
  Day 21 | 2.0 [1.6 to 2.5] | 2.4 [1.9 to 2.9]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.5 [1.2 to 1.8] | 1.4 [1.2 to 1.7]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 7.1 [5.2 to 9.7] | 13.8 [9.6 to 19.8]

107. Primary Outcome: Percentage of Subjects With RG Reassortant Virus (H5N8) Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 99
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 100 [88.4 to 100]
  Day 21 | 100 [88.4 to 100]

108. Primary Outcome: RG Reassortant Virus (H5N8) Antibody Titers (by MN) - Adult FLU D-QIV-015 Cohort
Description: as for outcome 92
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Titer
  Day 0 | 18.7 [16.8 to 20.7]
  Day 21 | 22.4 [20.4 to 24.8]

109. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for RG Reassortant Virus (H5N8) Antibody Titer by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 97
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects | 0.0 [0.0 to 11.6]

110. Primary Outcome: Mean Geometric Increase (MGI) for RG Reassortant Virus (H5N8) Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 94
Time Frame: At D21 (post-dose1 compared to D0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Ratio | 1.2 [1.1 to 1.4]

111. Primary Outcome: Percentage of Subjects With H1N1 Swine Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/Dilution ).
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 28 | 29 | 30
Percentage of subjects
  Day 0: number analyzed (Participants) | 28 | 27 | 29
  Day 0 | 100 [87.7 to 100] | 96.3 [81.0 to 99.9] | 96.6 [82.2 to 99.9]
  Day 42: number analyzed (Participants) | 25 | 29 | 30
  Day 42 | 100 [86.3 to 100] | 93.1 [77.2 to 99.2] | 100 [88.4 to 100]

112. Primary Outcome: H1N1 Swine Flu Virus Antibody Titers (by MN) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, Geometric mean titers (GMTs) were calculated with 95% CI for each treatment group within each study cohort.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 28 | 29 | 30
Titer
  Day 0: number analyzed (Participants) | 28 | 27 | 29
  Day 0 | 15.6 [12.5 to 19.5] | 24.6 [15.9 to 38.0] | 24.8 [17.7 to 34.8]
  Day 42: number analyzed (Participants) | 25 | 29 | 30
  Day 42 | 338.2 [257.5 to 444.4] | 78.1 [48.6 to 125.6] | 87.7 [65.9 to 116.8]

113. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1 Swine Flu Virus Antibody Titer by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination. seropositive subjects = titer ≥ 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 24 | 27 | 29
Percentage of subjects | 95.8 [78.9 to 99.9] | 55.6 [35.3 to 74.5] | 55.2 [35.7 to 73.6]

114. Primary Outcome: Mean Geometric Increase (MGI) for H1N1 Swine Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMT over pre-vaccination GMT.
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 24 | 27 | 29
Ratio | 21.4 [14.7 to 31.1] | 3.0 [1.6 to 5.7] | 3.4 [2.5 to 4.6]

115. Primary Outcome: Percentage of Subjects With H1N1 Swine Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titerss greater or equal than 10 1/DIL.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects
  Day 0 | 100 [89.4 to 100]
  Day 42 | 100 [89.4 to 100]

116. Primary Outcome: H1N1 Swine Flu Virus Antibody Titers (by MN) -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 112
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Titer
  Day 0 | 18.8 [13.3 to 26.5]
  Day 42 | 62.2 [40.0 to 96.8]

117. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1 Swine Flu Virus Antibody Titer by MN - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Percentage of subjects | 51.5 [33.5 to 69.2]

118. Primary Outcome: Mean Geometric Increase (MGI) for H1N1 Swine Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines
Description: as for outcome 114
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Ratio | 3.3 [2.3 to 4.7]

119. Primary Outcome: Percentage of Subjects With H1N1 Swine Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/DIL.
Time Frame: as for outcome 99
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 100 [86.8 to 100] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 100 [86.8 to 100] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 100 [88.1 to 100]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 100 [87.7 to 100]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 100 [86.3 to 100] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]

120. Primary Outcome: H1N1 Swine Flu Virus Enzyme-linked Immunosorbent Assay (ELISA) Antibody Titers - Adult Q-PAN-005 Cohort
Description: as for outcome 112
Time Frame: as for outcome 99
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Titer
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 20.5 [15.5 to 27.2] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 68.2 [42.0 to 110.6] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 19.1 [14.7 to 24.8]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 78.0 [53.2 to 114.5]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 42.3 [29.2 to 61.1] | 47.2 [30.9 to 72.0]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 84.8 [57.7 to 124.6] | 77.3 [55.9 to 106.8]

121. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1 Swine Flu Virus Antibody Titer by MN - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1 swine Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination. seropositive subjects = titer ≥ 10 1/DIL for H1N1 swine Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 65.4 [44.3 to 82.8] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 57.1 [37.2 to 75.5]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 62.5 [40.6 to 81.2] | 50.0 [27.2 to 72.8]

122. Primary Outcome: Mean Geometric Increase (MGI) for H1N1 Swine Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 114
Time Frame: as for outcome 102
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 3.3 [2.0 to 5.5] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 4.0 [2.5 to 6.4]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 2.1 [1.4 to 2.9] | 2.1 [1.5 to 3.1]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 4.0 [2.7 to 5.9] | 3.6 [2.3 to 5.7]

123. Primary Outcome: Percentage of Subjects With H1N1 Swine Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult H5N1-012 Cohort
Description: as for outcome 119
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Percentage of subjects
  Day 0 | 100 [93.3 to 100] | 98.0 [89.1 to 99.9]
  Day 21: number analyzed (Participants) | 53 | 47
  Day 21 | 100 [93.3 to 100] | 97.9 [88.7 to 99.9]
  Month 12 + 21 Days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 Days | 100 [92.6 to 100] | 100 [92.5 to 100]

124. Primary Outcome: H1N1 Swine Flu Virus Antibody Titers (by MN) - Adult H5N1-012 Cohort
Description: as for outcome 112
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 49
Titer
  Day 0 | 20.0 [15.9 to 25.2] | 18.4 [14.4 to 23.4]
  Day 21: number analyzed (Participants) | 53 | 47
  Day 21 | 75.9 [59.9 to 96.2] | 94.1 [68.4 to 129.3]
  Month 12 + 21 Days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 Days | 73.4 [55.4 to 97.1] | 72.2 [55.4 to 94.0]

125. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1 Swine Flu Virus Antibody Titer by MN - Adult H5N1-012 Cohort
Description: as for outcome 121
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 47
Percentage of subjects
  Day 21 | 64.2 [49.8 to 76.9] | 70.2 [55.1 to 82.7]
  Month 12 + 21 Days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 Days | 52.1 [37.2 to 66.7] | 55.3 [40.1 to 69.8]

126. Primary Outcome: Mean Geometric Increase (MGI) for H1N1 Swine Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult H5N1-012 Cohort
Description: as for outcome 114
Time Frame: At D21 (post-dose[ps-d]1), M12 (ps-d1) and M12+21days (ps-d2) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 48
Ratio
  Day 21: number analyzed (Participants) | 53 | 47
  Day 21 | 3.8 [2.8 to 5.1] | 5.2 [3.9 to 7.0]
  Month 12: number analyzed (Participants) | 50 | 48
  Month 12 | 1.3 [1.0 to 1.7] | 1.9 [1.5 to 2.5]
  Month 12 + 21 Days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 Days | 3.4 [2.5 to 4.7] | 4.2 [3.1 to 5.7]

127. Primary Outcome: Percentage of Subjects With H1N1 Swine Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 119
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- DQIV_NAS: Subjects 18-≤39 years of age (in D-QIVcohort of primary completed study FLU D-QIV-015 (201251) (A/Christchurch/16/2010 (H1N1)pdm09, A/Texas/50/2012 (H3N2), B/Massachusetts/02/2012, B/Brisbane/60/2008)) who were administered 15 µg HA (no AS) of each of 4 strains (total 60 µg HA) at Day 0.
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Percentage of subjects
  Day 0 | 96.7 [82.8 to 99.9]
  Day 21: number analyzed (Participants) | 28
  Day 21 | 100 [87.7 to 100]

128. Primary Outcome: H1N1 Swine Flu Virus Antibody Titers (by MN) - Adult FLU D-QIV-015 Cohort
Description: as for outcome 112
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 30
Titer
  Day 0 | 28.3 [19.8 to 40.5]
  Day 21: number analyzed (Participants) | 28
  Day 21 | 118.9 [88.4 to 159.9]

129. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1 Swine Flu Virus Antibody Titer by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 117
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 28
Percentage of subjects | 57.1 [37.2 to 75.5]

130. Primary Outcome: Mean Geometric Increase (MGI) for H1N1 Swine Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 114
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 28
Ratio | 4.3 [2.8 to 6.6]

131. Primary Outcome: Percentage of Subjects With H1N1pdm09-like Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/Dilution).
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 21 | 23 | 30
Percentage of subjects
  Day 0: number analyzed (Participants) | 21 | 20 | 29
  Day 0 | 100 [83.9 to 100] | 100 [83.2 to 100] | 100 [88.1 to 100]
  Day 42: number analyzed (Participants) | 18 | 23 | 30
  Day 42 | 100 [81.5 to 100] | 100 [85.2 to 100] | 100 [88.4 to 100]

132. Primary Outcome: H1N1pdm09-like Flu Virus Antibody Titers (by MN) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, Geometric mean titers (GMTs) were calculated with 95% CI for each treatment group within each study cohort.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 21 | 23 | 30
Titer
  Day 0: number analyzed (Participants) | 21 | 20 | 29
  Day 0 | 17.5 [12.9 to 23.9] | 25.5 [14.9 to 43.7] | 41.0 [27.2 to 61.6]
  Day 42: number analyzed (Participants) | 18 | 23 | 30
  Day 42 | 186.6 [120.8 to 288.4] | 52.5 [37.5 to 73.3] | 60.6 [43.6 to 84.3]

133. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1pdm09-like Flu Virus Antibody Titer by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination. seropositive subjects = titer ≥ 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 13 | 19 | 29
Percentage of subjects | 84.6 [54.6 to 98.1] | 42.1 [20.3 to 66.5] | 6.9 [0.8 to 22.8]

134. Primary Outcome: Mean Geometric Increase (MGI) for H1N1pdm09-like Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Mean Geometric Increase (MGI) = post-vaccination GMT over pre-vaccination GMT.
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H1N1_AS | H5N1_AS | H9N2_AS
Number analyzed (Participants) | 13 | 19 | 29
Ratio | 9.9 [5.7 to 17.2] | 1.9 [1.1 to 3.4] | 1.4 [1.2 to 1.8]

135. Primary Outcome: Percentage of Subjects With H1N1pdm09-like Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titerss greater or equal than 10 1/DIL.
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 32
Percentage of subjects
  Day 0: number analyzed (Participants) | 30
  Day 0 | 100 [88.4 to 100]
  Day 42 | 100 [89.1 to 100]

136. Primary Outcome: H1N1pdm09-like Flu Virus Antibody Titers (by MN) -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 132
Time Frame: At Day 0 (Pre-vaccination), Day 42 (Post-vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 32
Titer
  Day 0: number analyzed (Participants) | 30
  Day 0 | 40.9 [22.9 to 73.0]
  Day 42 | 56.6 [31.0 to 103.3]

137. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1pdm09-like Flu Virus Antibody Titer by MN - Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer.
Time Frame: At Day 42 (post-vaccination2 compared to pre-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 30
Percentage of subjects | 3.3 [0.1 to 17.2]

138. Primary Outcome: Mean Geometric Increase (MGI) for H1N1pdm09-like Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN -Pediatric Q-PAN H5N1-AS03-021 Cohort (Only AS Vaccines)
Description: as for outcome 134
Time Frame: At Day 42 (post-vaccination2/ pre-vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 30
Ratio | 1.3 [1.1 to 1.6]

139. Primary Outcome: Percentage of Subjects With H1N1pdm09-like Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. Seropositivity rate was defined as the percentage of subjects with titers greater or equal than 10 1/DIL.
Time Frame: as for outcome 99
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Percentage of subjects
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 92.3 [74.9 to 99.1] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 96.2 [80.4 to 99.9] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 89.7 [72.6 to 97.8]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 96.4 [81.7 to 99.9]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 96.0 [79.6 to 99.9] | 100 [83.9 to 100]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 100 [85.8 to 100] | 100 [83.2 to 100]

140. Primary Outcome: H1N1pdm09-like Flu Virus Enzyme-linked Immunosorbent Assay (ELISA) Antibody Titers - Adult Q-PAN-005 Cohort
Description: as for outcome 132
Time Frame: as for outcome 99
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 29
Titer
  Day 0: number analyzed (Participants) | 26 | 0
  Day 0 | 12.4 [9.5 to 16.1] |
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 19.0 [14.3 to 25.2] |
  Day 182: number analyzed (Participants) | 0 | 29
  Day 182 |  | 12.4 [9.6 to 16.0]
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 24.4 [17.9 to 33.2]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 22.3 [15.2 to 32.8] | 26.9 [17.7 to 40.9]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 33.6 [22.8 to 49.6] | 31.4 [20.8 to 47.4]

141. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1pdm09-like Flu Virus Antibody Titer by MN - Adult Q-PAN-005 Cohort
Description: With respect to samples from HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and quadrivalent inactivated seasonal, influenza vaccines, analysis was performed for measuring levels of H1N1pdm09-like Flu virus antibody by MN for all subjects who received an AS vaccine in each study cohort, aggregate variables were calculated with 95% CI for each treatment group within each study cohort. seronegative subjects = titer < 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination seropositive subjects = titer ≥ 10 1/DIL for H1N1pdm09-like Flu virus MN prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody titer ≥ 20 1/DIL at post-vaccination; For initially seropositive subjects, antibody titer at post-vaccination ≥ 4-fold the pre-vaccination antibody titer. The ≥4-fold increases were only calculated relative to baseline.
Time Frame: as for outcome 38
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Percentage of subjects
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 15.4 [4.4 to 34.9] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 25.0 [10.7 to 44.9]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 25.0 [9.8 to 46.7] | 35.0 [15.4 to 59.2]

142. Primary Outcome: Mean Geometric Increase (MGI) for H1N1pdm09-like Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination - Adult Q-PAN-005 Cohort
Description: as for outcome 134
Time Frame: as for outcome 102
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | QPAN5_C | QPAN5_G
Number analyzed (Participants) | 26 | 28
Ratio
  Day 42: number analyzed (Participants) | 26 | 0
  Day 42 | 1.5 [1.2 to 2.0] |
  Day 224: number analyzed (Participants) | 0 | 28
  Day 224 |  | 1.9 [1.5 to 2.5]
  Day 549: number analyzed (Participants) | 25 | 21
  Day 549 | 1.8 [1.3 to 2.5] | 2.0 [1.5 to 2.7]
  Day 591: number analyzed (Participants) | 24 | 20
  Day 591 | 2.6 [1.8 to 3.7] | 2.2 [1.6 to 3.0]

143. Primary Outcome: Percentage of Subjects With H1N1pdm09-like Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult H5N1-012 Cohort
Description: as for outcome 139
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 48
Percentage of subjects
  Day 0 | 96.2 [87.0 to 99.5] | 97.9 [88.9 to 99.9]
  Day 21: number analyzed (Participants) | 53 | 46
  Day 21 | 100 [93.3 to 100] | 100 [92.3 to 100]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 97.9 [88.9 to 99.9] | 97.9 [88.7 to 99.9]

144. Primary Outcome: H1N1pdm09-like Flu Virus Antibody Titers (by MN) - Adult H5N1-012 Cohort
Description: as for outcome 132
Time Frame: At D0 (Pre), D21 (Post-dose 1) and M12+21days (post-dose2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 48
Titer
  Day 0 | 11.9 [10.7 to 13.2] | 13.7 [11.1 to 17.0]
  Day 21: number analyzed (Participants) | 53 | 46
  Day 21 | 22.8 [19.1 to 27.2] | 27.0 [22.1 to 33.1]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 47
  Month 12 + 21 days | 21.2 [17.4 to 25.8] | 23.2 [19.2 to 28.0]

145. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1pdm09-like Flu Virus Antibody Titer by MN - Adult H5N1-012 Cohort
Description: as for outcome 141
Time Frame: At D21 (post-dose1 compared to [/]D0), at M12+21days (post-dose2 /D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 46
Percentage of subjects
  Day 21: number analyzed (Participants) | 53 | 45
  Day 21 | 18.9 [9.4 to 32.0] | 26.7 [14.6 to 41.9]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 46
  Month 12 + 21 days | 22.9 [12.0 to 37.3] | 21.7 [10.9 to 36.4]

146. Primary Outcome: Mean Geometric Increase (MGI) for H1N1pdm09-like Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult H5N1-012 Cohort
Description: as for outcome 134
Time Frame: At D21 (post-dose[ps-d]1), M12 (ps-d1) and M12+21days (ps-d2) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 53 | 47
Ratio
  Day 21: number analyzed (Participants) | 53 | 45
  Day 21 | 1.9 [1.6 to 2.3] | 2.1 [1.6 to 2.7]
  Month 12: number analyzed (Participants) | 50 | 47
  Month 12 | 1.2 [1.1 to 1.5] | 1.3 [1.0 to 1.6]
  Month 12 + 21 days: number analyzed (Participants) | 48 | 46
  Month 12 + 21 days | 1.8 [1.5 to 2.2] | 1.7 [1.3 to 2.2]

147. Primary Outcome: Percentage of Subjects With H1N1pdm09-like Flu Virus Antibody Titer (by MN) Equal or Above the Cut-off of 10 1/DIL - Adult FLU D-QIV-015 Cohort
Description: as for outcome 139
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 29
Percentage of subjects
  Day 0 | 96.6 [82.2 to 99.9]
  Day 21: number analyzed (Participants) | 28
  Day 21 | 100 [87.7 to 100]

148. Primary Outcome: H1N1pdm09-like Flu Virus Antibody Titers (by MN) - Adult FLU D-QIV-015 Cohort
Description: as for outcome 132
Time Frame: At D0 (Pre), D21 (Post-dose 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 29
Titer
  Day 0 | 38.1 [25.6 to 56.8]
  Day 21: number analyzed (Participants) | 28
  Day 21 | 312.2 [215.8 to 451.6]

149. Primary Outcome: Percentage of Subjects With a ≥4-fold Rise for H1N1pdm09-like Flu Virus Antibody Titer by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 137
Time Frame: At D21 (post-dose1 compared to [/]D0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 27
Percentage of subjects | 77.8 [57.7 to 91.4]

150. Primary Outcome: Mean Geometric Increase (MGI) for H1N1pdm09-like Flu Virus Antibody Post-vaccination Concentration Compared to Pre-vaccination, by MN - Adult FLU D-QIV-015 Cohort
Description: as for outcome 134
Time Frame: At D21 (post-dose1) compared to D0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DQIV_NAS
Number analyzed (Participants) | 27
Ratio | 8.2 [5.0 to 13.6]

151. Secondary Outcome: GMCs of Anti-H1 HA Stalk ELISA Antibody - Adult Q-PAN H1N1-019 Cohort
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all the subjects in the adult CCPan H5N1-001, the Q-Pan H1N1-019 and the Q-Pan H9N2-001 study cohorts. Geometric mean concentration (AS Group and no AS group within each study) was calculated with 95% CI at each specified time point and expressed in Elisa Unit per milliliter (EU/mL).
Time Frame: At D21, D42, and D182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H1N1_AS | H1N1_NAS
Number analyzed (Participants) | 29 | 29
EU/mL
  Day 21: number analyzed (Participants) | 28 | 25
  Day 21 | 45098.3 [34775.1 to 58486.2] | 37969.9 [26930.8 to 53534.1]
  Day 42: number analyzed (Participants) | 27 | 27
  Day 42 | 46177.1 [37510.4 to 56846.2] | 38598.2 [27818.0 to 53555.9]
  Day 182 | 21782.4 [17803.2 to 26651.0] | 24705.6 [18369.2 to 33227.7]
Statistical Analysis 1: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H1N1_AS over H1N1_NAS) at Day 21. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; ANCOVA model on logarithm10 transformation of concentration, with vaccine group as fixed effect and anti- H1 stalk ELISA result at Day 0 as covariates; Adjusted GMC ratio = 1.12, 95% CI 2-sided [0.73 to 1.72]
Statistical Analysis 2: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H1N1_AS over H1N1_NAS) at Day 42. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.23, 95% CI 2-sided [0.83 to 1.81]
Statistical Analysis 3: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H1N1_AS over H1N1_NAS) at Day 182. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 0.88, 95% CI 2-sided [0.63 to 1.24]

152. Secondary Outcome: GMCs of Anti-H1 HA Stalk ELISA Antibody - Adult CC-PAN H5N1-001 Cohort
Description: as for outcome 151
Time Frame: At D21, D42, D182 and Day 385
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H5N1_AS | H5N1_NAS
Number analyzed (Participants) | 29 | 27
EU/mL
  Day 21 | 46013.8 [33592.9 to 63027.5] | 27845.9 [20269.3 to 38254.5]
  Day 42 | 68348.8 [53244.4 to 87738.1] | 31718.0 [23755.4 to 42349.5]
  Day 182 | 33610.2 [26464.5 to 42685.3] | 17401.9 [13330.1 to 22717.5]
  Day 385 | 25346.9 [20205.0 to 31797.3] | 15768.2 [11999.3 to 20720.9]
Statistical Analysis 1: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H5N1_AS over H5N1_NAS) at Day 21 . Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.66, 95% CI 2-sided [1.12 to 2.47]
Statistical Analysis 2: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H5N1_AS over H5N1_NAS) at Day 42. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 2.16, 95% CI 2-sided [1.54 to 3.03]
Statistical Analysis 3: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H5N1_AS over H5N1_NAS) at Day 182. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.95, 95% CI 2-sided [1.49 to 2.54]
Statistical Analysis 4: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H5N1_AS over H5N1_NAS) at Day 385 . Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.63, 95% CI 2-sided [1.32 to 2.01]

153. Secondary Outcome: GMCs of Anti-H1 HA Stalk ELISA Antibody - Adult Q-PAN H9N2-001 Cohort
Description: as for outcome 151
Time Frame: At D21, D42 and D182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 30 | 30
EU/mL
  Day 21 | 25189.3 [20983.6 to 30238.0] | 16592.8 [13332.5 to 20650.4]
  Day 42 | 31665.4 [27405.9 to 36587.0] | 19681.1 [16293.6 to 23772.7]
  Day 182: number analyzed (Participants) | 28 | 30
  Day 182 | 20570.2 [16717.6 to 25310.5] | 15471.1 [11913.9 to 20090.4]
Statistical Analysis 1: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H9N2_AS over H9N2_NAS) at Day 21. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.39, 95% CI 2-sided [1.14 to 1.69]
Statistical Analysis 2: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H9N2_AS over H9N2_NAS) at Day 42. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.49, 95% CI 2-sided [1.28 to 1.73]
Statistical Analysis 3: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Adjusted GMC ratios of anti-H1 HA stalk ELISA antibody concentration between groups (H9N2_AS over H9N2_NAS) at Day 182. Adjusted GMC = GMC adjusted for baseline concentration; ANCOVA; [statistical method as in outcome 151, analysis 1]; Adjusted GMC ratio = 1.20, 95% CI 2-sided [1.00 to 1.44]

154. Secondary Outcome: Percentage of Subjects With at Least 4-fold Increase of Anti-H1 Stalk ELISA - Adult Q-PAN H1N1-019 Cohort
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1,and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring levels of anti-H1 stalk antibody by ELISA for all the subjects in the adult CCPan H5N1-001, the Q-Pan H1N1-019 and the Q-Pan H9N2-001 study cohorts. Percentage of subjects with at least 4-fold increase to anti-H1 stalk ELISA was calculated with 95% CI at each specified time point. seronegative subjects = concentration < 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. seropositive subjects = concentration ≥ 66 EU/mL for anti-H1 stalk ELISA prior to vaccination. 4-fold increase defined as: For initially seronegative subjects, antibody concentration ≥ 132 EU/mL at post-vaccination. For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: At D21, D42, and D182 (compared to Day 0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H1N1_AS | H1N1_NAS
Number analyzed (Participants) | 27 | 25
Percentage of subjects
  Day 21: number analyzed (Participants) | 27 | 23
  Day 21 | 63.0 [42.4 to 80.6] | 52.2 [30.6 to 73.2]
  Day 42: number analyzed (Participants) | 25 | 25
  Day 42 | 72.0 [50.6 to 87.9] | 60.0 [38.7 to 78.9]
  Day 182 | 25.9 [11.1 to 46.3] | 32.0 [14.9 to 53.5]
Statistical Analysis 1: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Difference between groups (H1N1_AS minus H1N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 21; Asymptotic standardized 95% CI; Difference in percentage of subjects = 10.79, 95% CI 2-sided [-16.50 to 36.83]
Statistical Analysis 2: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Difference between groups (H1N1_AS minus H1N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 42; Asymptotic standardized 95% CI; Difference in percentage of subjects = 12.00, 95% CI 2-sided [-14.45 to 36.98]
Statistical Analysis 3: Comparison: H1N1_AS vs H1N1_NAS; Test type: Equivalence — Difference between groups (H1N1_AS minus H1N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 182; Asymptotic standardized 95% CI; Difference in percentage of subjects = -6.07, 95% CI 2-sided [-30.56 to 18.65]

155. Secondary Outcome: Percentage of Subjects With at Least 4-fold Increase of Anti-H1 Stalk ELISA - Adult CC-PAN H5N1-001 Cohort
Description: as for outcome 154
Time Frame: At D21, D42, D182 and Day 385 (compared to Day 0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H5N1_AS | H5N1_NAS
Number analyzed (Participants) | 29 | 27
Percentage of subjects
  Day 21 | 34.5 [17.9 to 54.3] | 7.4 [0.9 to 24.3]
  Day 42 | 55.2 [35.7 to 73.6] | 18.5 [6.3 to 38.1]
  Day 182 | 13.8 [3.9 to 31.7] | 7.4 [0.9 to 24.3]
  Day 385 | 6.9 [0.8 to 22.8] | 0.0 [0.0 to 12.8]
Statistical Analysis 1: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Difference between groups (H5N1_AS minus H5N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 21; Asymptotic standardized 95% CI; Difference in percentage of subjects = 27.08, 95% CI 2-sided [5.96 to 47.01]
Statistical Analysis 2: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Difference between groups (H5N1_AS minus H5N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 42; Asymptotic standardized 95% CI; Difference in percentage of subjects = 36.65, 95% CI 2-sided [11.41 to 57.53]
Statistical Analysis 3: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Difference between groups (H5N1_AS minus H5N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 182; Asymptotic standardized 95% CI; Difference in percentage of subjects = 6.39, 95% CI 2-sided [-11.91 to 24.71]
Statistical Analysis 4: Comparison: H5N1_AS vs H5N1_NAS; Test type: Equivalence — Difference between groups (H5N1_AS minus H5N1_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 365; Asymptotic standardized 95% CI; Difference in percentage of subjects = 6.90, 95% CI 2-sided [-6.19 to 22.15]

156. Secondary Outcome: Percentage of Subjects With at Least 4-fold Increase of Anti-H1 Stalk ELISA - Adult Q-PAN H9N2-001 Cohort
Description: as for outcome 154
Time Frame: At D21, D42 and D182 (compared to Day 0)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 30 | 30
Percentage of subjects
  Day 21 | 10.0 [2.1 to 26.5] | 6.7 [0.8 to 22.1]
  Day 42 | 20.0 [7.7 to 38.6] | 3.3 [0.1 to 17.2]
  Day 182: number analyzed (Participants) | 28 | 30
  Day 182 | 3.6 [0.1 to 18.3] | 3.3 [0.1 to 17.2]
Statistical Analysis 1: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Difference between groups (H9N2_AS minus H9N2_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 21; Asymptotic standardized 95% CI; Difference in percentage of subjects = 3.33, 95% CI 2-sided [-13.06 to 20.24]
Statistical Analysis 2: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Difference between groups (H9N2_AS minus H9N2_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 42; Asymptotic standardized 95% CI; Difference in percentage of subjects = 16.67, 95% CI 2-sided [0.35 to 34.76]
Statistical Analysis 3: Comparison: H9N2_AS vs H9N2_NAS; Test type: Equivalence — Difference between groups (H9N2_AS minus H9N2_NAS) in percentage of subjects with at least 4-fold increase of anti-H1 stalk ELISA at Day 182; Asymptotic standardized 95% CI; Difference in percentage of subjects = 0.24, 95% CI 2-sided [-13.76 to 15.00]

157. Secondary Outcome: Number of Subjects With Seropositivity Status at Baseline (Day 0) for the HI Assay Against the Pandemic Vaccine Homologous Virus - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 Cohorts
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1, and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring the number of subjects with seropositivity status at baseline (Day 0) for the HI assay against the pandemic vaccine homologous virus - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001 cohorts. Seronegative subjects = Subjects with antibody titer < 10 1/DIL for Pandemic vaccine homologous virus and Seropositive subjects = Subjects with antibody titer ≥ 10 1/DIL for Pandemic vaccine homologous virus (i.e., A/California/7/2009 for subjects from the Q-PAN H1N1-019 study, A/Indonesia/5/2005 for subjects from CC-PAN H5N1-001 study, A/chicken/Hong Kong/G9/1997 for subjects from Q-PAN H9N2-001 study).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30
Participants
  Seronegative | 17 | 19 | 20 | 26 | 19 | 18
  Seropositive | 12 | 10 | 9 | 1 | 11 | 12

158. Secondary Outcome: Number of Subjects With Seropositivity Status at Pre-vaccination (Baseline) for the HI Assay Against the Pandemic Vaccine Homologous Virus - Adult FLU D-QIV-015, Q-PAN-005, H5N1-012 Cohorts
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1, and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring the number of subjects with seropositivity status at baseline (at Day 0 in all subjects except for group G of Q-PAN-005 [i.e, at Day182]) for the HI assay against the pandemic vaccine homologous virus - Adult FLU D-QIV-015, Q-PAN-005, H5N1-012 cohorts . Seronegative subjects = Subjects with antibody titer < 10 1/DIL for Pandemic vaccine homologous virus and Seropositive subjects = Subjects with antibody titer ≥ 10 1/DIL for Pandemic vaccine homologous virus (i.e., for FLU D-QIV-015: A/Christchurch/16/2010 at Day 0, for Q-PAN-005 study, group C: A/Turkey/01/2005 and A/Indonesia/5/2005 at Day 0 and for group G, A/Turkey/01/2005 at Day 182, for H5N1-012 study, for group VT/VT/12M : A/Vietnam/1194/2004 at Day 0, for group VT/IN/12M, A/Indonesia/5/2005 and A/Vietnam/1194/2004-like at Day 0).
Time Frame: At Day 0, (except for group G of Q-PAN-005, at Day182)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DQIV_NAS | QPAN5_C | QPAN5_G | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 30 | 26 | 29 | 53 | 49
Participants
  A/Christchurch/16/2010-seronegative | 3 | 0 | 0 | 0 | 0
  A/Christchurch/16/2010-seropositive | 27 | 0 | 0 | 0 | 0
  A/Christchurch/16/2010-missing | 0 | 26 | 29 | 53 | 49
  A/Indonesia/5/2005-seronegative | 0 | 26 | 0 | 0 | 49
  A/Indonesia/5/2005-seropositive | 0 | 0 | 0 | 0 | 0
  A/Indonesia/5/2005-missing | 30 | 0 | 29 | 53 | 0
  A/Turkey/01/2005-seronegative | 0 | 25 | 24 | 0 | 0
  A/Turkey/01/2005-seropositive | 0 | 1 | 5 | 0 | 0
  A/Turkey/01/2005-missing | 30 | 0 | 0 | 53 | 49
  A/Vietnam/1194/2004-like-seronegative | 0 | 0 | 0 | 52 | 49
  A/Vietnam/1194/2004-like-seropositive | 0 | 0 | 0 | 1 | 0
  A/Vietnam/1194/2004-like-missing | 30 | 26 | 29 | 0 | 0

159. Secondary Outcome: Number of Subjects With Seropositivity Status at Pre-vaccination (Baseline) for the HI Assay Against A/California/7/09 Virus (or Like Virus) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001, Q-PAN-005, H5N1-012 Cohorts
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1, and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring the number of subjects with seropositivity status at pre-vaccination (Baseline) for the HI assay against A/California/7/09 virus (or like virus) - Adult Q-PAN H1N1-019, CC-PAN H5N1-001, Q-PAN H9N2-001, Q-PAN-005, H5N1-012 cohorts. Seronegative subjects = Subjects with antibody titer < 10 1/DIL for A/California/7/09 virus (or like virus) and Seropositive subjects = Subjects with antibody titer ≥ 10 1/DIL for A/California/7/09 virus (or like virus).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS | QPAN5_C | QPAN5_G | H5N1_VT | H5N1_IN
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 30 | 30 | 26 | 29 | 53 | 49
Participants
  Seronegative | 17 | 19 | 7 | 9 | 4 | 7 | 16 | 15 | 31 | 32
  Seropositive | 12 | 10 | 21 | 18 | 26 | 23 | 10 | 14 | 19 | 15
  Missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2

160. Secondary Outcome: Number of Subjects With Seropositivity Status Against Flu A/Indonesia/05/2005 (H5N1) HI Antibodies - Pediatric H5N1 Cohort
Description: With respect to samples from the HA Group 1-related studies (i.e., with H1N1, H5N1, and H9N2 pandemic, and IIV4 seasonal, influenza vaccines), analysis was performed for measuring the number of subjects with seropositivity status against Flu A/Indonesia/05/2005 (H5N1) HI antibodies - Pediatric H5N1 cohort. Seronegative subjects = Subjects with antibody titer < 10 1/DIL for Flu A/Ind/05/05 (H5N1).HA HI prior to vaccination and Seropositive subjects = Subjects with antibody titer ≥ 10 1/DIL for Flu A/Ind/05/05 (H5N1).HA HI prior to vaccination.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1_PAS
Number analyzed (Participants) | 33
Participants | 33

ADVERSE EVENTS:
Time Frame: Not applicable since subjects were enrolled in the primary studies and there was no enrollment in that study. Therefore, safety was not assessed in this study.
Description: Not applicable since subjects were enrolled in the primary studies and there was no enrollment in that study. Therefore, safety was not assessed in this study.
Arm/Group | H1N1_AS | H1N1_NAS | H5N1_AS | H5N1_NAS | H9N2_AS | H9N2_NAS | DQIV_NAS | QPAN5_C | QPAN5_G | H5N1_VT | H5N1_IN | H5N1_PAS | H5N1_PCN
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02415842/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02415842/SAP_001.pdf